CLINICAL TRIAL: NCT05742945
Title: Can Immediate Lymphatic Reconstruction With Lymphatico-Venous Anastomosis Reduce the Occurrence of Arm Lymphedema in Breast Cancer Patients After Axillary Lymph Node Dissection? A Prospective Randomized Controlled Trial.
Brief Title: Can ILR Reduce the Risk of Arm Lymphedema?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202207198RINB
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ILR (Experimental): Breast cancer patients receiving axillary lymph node dissection and immediate lymphatic reconstruction
  Interventions: Procedure: Immediate lymphatic reconstruction
- non-ILR (No Intervention): Breast cancer patients receiving only axillary lymph node dissection

INTERVENTIONS:
Procedure: Immediate lymphatic reconstruction — Breast cancer patients receive axillary lymph node dissection and immediate lymphatic reconstruction
  Arms: ILR

SUMMARY:
Breast cancer-related lymphedema (BCRL) is a debilitating, usually lifelong burden for breast cancer survivors. For the breast cancer patients receiving axillary lymph node dissection (ALND), the likelihood of BCRL is about 20%. Lymphatico-venous anastomosis (LVA) has been accepted as a method of treating extremity lymphedema. A few studies have mentioned the prophylactic effect of LVA on BCRL. However, there is still lack of a large-scale randomized controlled trial to corroborate its efficacy. Therefore, the goal of this study is to conduct a prospective randomized controlled trial to evaluate if immediate lymphatic reconstruction (ILR) with LVA could have a clinically significant effect on the reduction of BCRL occurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with unilateral breast cancer
2. Going to receive axillary lymph node dissection, or sentinel lymph node biopsy but being highly suspected of axillary metastasis preoperatively

Exclusion Criteria:

1. Had received axillary lymph node dissection
2. Going to receive bilateral axillary lymph node dissections
3. Already have arm lymphedema
4. Allergy to the dye used intraoperatively

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Arm lymphedema | Two years
  Occurrence of arm lymphedema

SECONDARY OUTCOMES:
Drainage amount | Two weeks
  Drainage amount from operative wounds
Seroma or lymphocele | One month
  Occurrence of seroma or lymphocele
PROM | Two years
  Patient reported outcome measures by LYMPH-Q Upper Extremity Module
Subclinical lymphedema | Two years
  Occurrence of subclinical lymphedema

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Chih Dai, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Non-identifiable data will be shared upon request